

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

TAME: A pilot study of weekly paclitaxel, bevacizumab, and Tumor Associated Macrophage targeted therapy (zoledronic acid) in women with recurrent, platinum-resistant, Epithelial ovarian, fallopian tube or primary peritoneal cancer

| 2021 0001 | | |
|---|---|---|
| Subtitle: TAME | | WINDOWS CONTROL CONTRO |
| Study Chair: | Shannon N. V | Vestin, MD, MPH |
| Participant's Na | ime | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by the MD Anderson Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

2021-0694

The goal of this clinical research study is to learn if adding zoledronic acid to the combination of paclitaxel and bevacizumab can help control ovarian tube, fallopian tube, or primary peritoneal cancer that is relapsed (has come back) or refractory (has not responded to treatment).

<u>Please note</u>: If you take part in this study, you may be given either bevacizumab or a biosimilar of that drug (which means it is identical to the study drug). Everything stated in this document about bevacizumab also applies to its biosimilar, including information about FDA approval status, side effects, and cost.

This is an investigational study. Bevacizumab and paclitaxel are FDA approved and commercially available for the treatment of several types of cancer, including epithelial ovarian, primary peritoneal, and fallopian tube cancer. Zoledronic acid is FDA approved and commercially available for the treatment of bone complications in patients with multiple myeloma and patients with solid tumors. It is considered

investigational to give zoledronic acid with bevacizumab and paclitaxel to patients with relapsed/refractory ovarian tube, fallopian tube, or primary peritoneal cancer.

The study doctor can explain how the study drugs work.

The study drugs may help control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, such as possible side effects, potential costs, hospitalization, prolonged stay out of town, or other standard options available to you.

You can read a full list of potential side effects below in the Possible Risks section of this consent.

You may receive the study drugs for as long as the study doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Zoledronic acid will be provided at no cost to you during the study. You and/or your insurance provider will be responsible for the cost of bevacizumab and paclitaxel.

You may choose not to take part in this study. Instead of taking part in the study, you may choose to receive bevacizumab and paclitaxel. The study doctor will discuss the possible risks and benefits of these treatments. You may choose to receive other investigational therapy, if available. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

## 1. STUDY DETAILS

## **Screening Tests**

Signing this consent form does not meant that you will be able to part in this study. You will have the following screening tests within 28 days before starting your first dose of the study drugs to help the doctor decide if you are eligible:

- You will have a physical exam.
- You will have an EKG to check your heart function.
- Blood (about 5 tablespoons) will be drawn for routine tests and tests to check for hepatitis B, hepatitis C, and HIV (the AIDS virus). If you can become pregnant, part of this sample will be used for a pregnancy test. To take part in this study, you must not be pregnant.
- Urine will be collected for routine tests.
- You will have either a CT scan or MRI of the chest, abdomen, and pelvis to check the status of the disease.

- You will have a tissue biopsy to check the status of the disease. This sample
  will be compared to tissue samples collected later in the study to help
  researchers learn if the study drugs have affected the disease.
- If available and if less than 3 years old, leftover tumor tissue from a previously performed procedure will also be collected.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatments options will be discussed with you.

## Study Groups (Arms)

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to either Arm 1 or Arm 2:

- If you are in Arm 1, you will receive paclitaxel and bevacizumab.
- If you are in Arm 2, you will receive paclitaxel, bevacizumab, and zoledronic acid.

You will have an equal chance (50/50) of being assigned to either arm. This is done because no one knows if one arm is better, worse, or the same as the other. Both you and the study doctor will know which study drugs you are receiving.

Up to 30 participants (15 in each arm) will be enrolled in this study. All will take part at MD Anderson.

# Crossover Option (Arm 1)

If you are assigned to Arm 1 and the disease gets worse during the study, you may have the option to crossover to Arm 2 and begin receiving the study drugs with zoledronic acid. This option will be discussed with you.

## **Study Drug Administration**

Each study cycle is 28 days. You will receive the study drugs as follows:

- You will receive **paclitaxel** by vein over about 3 hours on Days 1, 8, and 15 of each cycle.
- You will receive **bevacizumab** by vein over about 60-90 minutes on Days 1 and 15 of each cycle.
- If you are in Arm 2, you will receive zoledronic acid by vein over about 30 minutes on Day 1 of each cycle.

If you are receiving bevacizumab and paclitaxel, you may choose to receive these 2 drugs at MD Anderson or at another hospital under the care of your home doctor. You may also choose to receive some of the study procedures described below (routine blood/urine tests and CT scans) outside of MD Anderson. The study doctor will discuss these options with you.

#### **Study Visits**

On Day 1 of every cycle:

- You will have a physical exam.
- Blood (about 5 tablespoons) will be drawn for routine and research tests and tests to check for biomarkers. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.
- During Cycles 1, 3, and 5, blood (about 5 teaspoons) will be drawn to check for a tumor marker called CA125 and for research testing related to how you respond to the study drugs. Tumor markers may be related to the status of the disease.
- Urine will be collected for routine tests.
- If you can become pregnant, part of the above blood/urine sample will be collected for a pregnancy test.

## On Days 8 and 15 of every cycle:

 Blood (about 5 tablespoons) will be drawn for routine and research tests and tests to check for biomarkers. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.

**Every 8 weeks**, you will have either a CT or MRI of the chest, abdomen, and pelvis to check the status of the disease.

After receiving the study drugs for about 2 cycles, you will have a tumor biopsy to compare to the tissue collected at screening for research testing related to your immune system and to learn if there have been any changes to the disease.

## **End of Treatment**

After you stop receiving the study drugs, the following tests and procedures will be performed:

- You will have a physical exam.
- Blood (about 5 tablespoons) will be drawn for routine and tumor marker testing.
   If you can become pregnant, part of this sample will be used for a pregnancy test.
- Urine will be collected for routine tests.

## **Follow-Up Visits**

About 30 days and 90 days after your last dose of study drugs:

- You will have a physical exam.
- Blood (about 5 tablespoons) will be drawn for routine tests. At the 90-day visit, this blood sample will also be used for research testing to check how you responded to the study drugs.
- Urine will be collected for routine tests.

If you stopped taking the study drugs because the disease got worse, you will come to the clinic every 12 weeks to have the above follow-up tests repeated.

If you stopped taking part in the study for reasons other than the disease getting worse or you do not want to come to the clinic every 12 weeks, you will be called by the

study staff every 6 months and asked how you are doing. This call should last about 5-10 minutes.

In all cases, follow-up will stop if you decide to leave the study, the study ends, or you want to join another research study or receive another type of anti-cancer treatment.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drug/procedures.

Bevacizumab, paclitaxel, and zoledronic acid each may cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become lifethreatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

## **Bevacizumab Side Effects**

# Common (occurring in more than 20% of patients)

- high blood pressure
- headache
- dizziness
- fatigue
- difficulty sleeping
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental
- high blood sugar (possible diabetes)
- weight loss
- loss of appetite
- diarrhea
- mouth blisters/sores (possible difficulty swallowing)
- nausea
- failure of the ovaries to produce hormones, which may be permanent (possible

- pain
- bleeding (including nosebleed)
- low blood cell counts (white, platelets)
- bleeding in the lungs and/or airways
- difficulty breathing
- cough
- infection

| status, and/or seizures) | stopped menstrual cycle) | |
|--------------------------|--------------------------|---|
| | | ! |

# Frequency Unknown but occurring in more than 10% of patients

| <ul> <li>shedding and<br/>the skin (poss<br/>loss of bodily)</li> </ul> | es |
|---|---|
|---|---|

## Occasional (occurring in 3-20% of patients)

- severe heart problems
- swelling (arm/leg)
- blood clots in a vein (possible pain, swelling, and/or redness)
- blood clots in an artery (possible organ damage such as stroke and/or heart attack)
- fainting
- anxiety
- difficulty forming or speaking words

- voice disorder
- wound healing problems after surgery
- abdominal pain
- dehydration
- constipation
- vein blockage in the abdomen
- hole in the intestines (possibly leaking contents into the abdomen)
- hemorrhoids
- pelvic pain

- abnormal kidney test (possible kidney damage)
- weakness (including muscle weakness)
- runny/stuffy nose
- infusion reaction (possible chills and/or hives)
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

Bevacizumab may occasionally cause an abnormal opening that develops between one area of the body and another (for example, an abnormal connection and opening in one or more places between the trachea [breathing tube] and esophagus, which may interfere with swallowing, digestion, and/or choking. Another example is abnormal connections or passageways between different parts of the digestive system and/or the vagina or rectum). These passageways or openings may also happen in the kidney or lungs. This may result in death.

## **Frequency Unknown**

| heart attack | temporary stroke | <ul> <li>vomiting up blood</li> </ul> |
|---|---|---|
| chest pain due to heart | symptoms | <ul> <li>vaginal bleeding</li> </ul> |
| trouble | <ul> <li>bleeding around the</li> </ul> | <ul> <li>coughing up blood</li> </ul> |
| • stroke | brain | <ul> <li>allergic reaction</li> </ul> |
| | digestive system | |
| | bleeding | |

## Rare but serious (occurring in fewer than 3% of patients)

- severe increase in blood pressure (possible stroke)
- weakness in wall of artery (possible serious bleeding complications)
- abnormal changes in the blood vessel that carries blood from the heart
- tear in a major blood vessel leading into the heart
- tearing of the walls around the heart
- brain injury that may be reversible (possible headache, confusion, seizures, and/or vision loss)
- decreased brain function due to high blood pressure

- decay of body tissue
- stomach and/or small intestine ulcer
- decreased blood flow to part of the bowel (possibly causing death of tissue)
- hole in the gall bladder (possible abdominal pain, gall stones, nausea, and/or infection)
- low red blood cell count
- bone destruction (including destruction of the jaw bone)
- inflammation inside the eye
- blurry vision
- deafness
- kidney failure

- abnormal blood clotting in small blood vessels of the kidney (possible kidney damage)
- increased blood pressure in the lungs (possible difficulty breathing and/or heart failure)
- blockage in the lung (possible pain, shortness of breath, and/or failure to breathe)
- abnormal hole inside the nose
- immune system response (possible loss of drug function)

Rarely (in about 1-2% of patients), bevacizumab may cause bleeding in the brain in patients who have received bevacizumab for the treatment of primary brain tumors. You will be monitored for this complication and removed from the study if this were to occur.

If you are taking Coumadin (warfarin) or other blood-thinning drugs, you may be at higher risk of blood clots and/or bleeding.

# **Paclitaxel Side Effects**

# Common (occurring in more than 20% of patients)

- abnormal EKG
- swelling
- flushing
- hair loss (partial or total)
- mouth blisters/sores (possible difficulty swallowing)
- nausea/vomiting
- diarrhea
- low blood cell counts (red/platelets/white)
- abnormal liver tests (possible liver damage)
- pain (muscle/joint)
- weakness

- nerve damage (possible numbness, pain, and/or loss of motor function)
- abnormal kidney test (possible kidney damage)
- wheezing/shortness of breath
- allergic reaction

| <ul> <li>infection</li> </ul> |
|-------------------------------|

# Occasional (occurring in 3-20% of patients)

- low blood pressure (possible dizziness/ fainting)
- slow heartbeat
- fever
- blood clots in a vein (possible pain, swelling, and/or redness)
- skin rash
- abdominal pain
- abnormal liver tests (possible yellowing of the skin and/or eyes)
- lung damage (possible shortness of breath)
- injection site reaction (possible redness, swelling, skin discoloration)

## Rare but serious (occurring in fewer than 3% of patients)

- fast/irregular heartbeat
- heart failure
- heart attack
- decreased blood supply to the heart
- high blood pressure
- fainting
- decreased brain function (possible paralysis and/or coma)
- decreased brain function due to liver damage
- seizure
- severe sunburn-like rash at site of previous radiation (called radiation recall)
- death of skin
- worsening of existing scleroderma (severe hardened skin, which can cause difficult movement)

- inflammation at the site of previous tissue death
- very severe blistering skin disease (with ulcers of the skin and digestive tract)
- very severe blistering skin disease (loss of large portion of skin)
- inflammation of the pancreas (possible abdominal pain)
- inflammation of the intestines
- dehydration
- hole in the intestines (possible leaking contents into the abdomen)
- decreased blood flow to part of the bowel (possibly causing death of tissue)
- paralysis of the intestines

- intestinal blockage
- difficulty walking
- liver damage and/or failure
- hearing loss
- decreased kidney function
- blockage in the lung (possible pain and/or shortness of breath)
- lung inflammation (possible difficulty breathing)
- blood clots in the lung (possible failure to breathe)
- difficulty breathing
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)
- tissue death at the injection site caused by drug leakage

# **Zoledronic Acid Side Effects**

Common (occurring in more than 20% of patients)

- swelling (legs/feet)
- fever
- fatigue
- nausea/vomiting
- constipation

- diarrhea
- loss of appetite
- low red blood cell count
- pain

- weakness
- kidney failure
- difficulty breathing
- cough

## Occasional (occurring in 3-20% of patients)

- low blood pressure (possible dizziness and/or fainting)
- chest pain
- headache
- dizziness
- sleepiness
- · difficulty sleeping
- anxiety
- depression
- agitation
- confusion
- numbness

- shivering
- hair loss (partial or total)
- skin rash
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- dehydration
- abdominal pain

- weight loss
- upset stomach
- difficulty swallowing
- sore throat
- mouth blisters/sores (possible difficulty swallowing)
- low blood cell count (white/platelets)
- abnormal sensation (such as pins and needles)
- worsening of cancer

# Rare but serious (occurring in fewer than 3% of patients)

- tissue swelling
- high blood pressure
- slow/irregular heartbeat
- seizure
- stroke
- very severe blistering skin disease (with ulcers of the skin and digestive tract)
- very severe blistering skin disease (loss of large portion of skin)
- high hormone blood levels resulting in high calcium blood levels (possible bone pain, nausea, and/or kidney stones)
- decreased kidney function (possible kidney failure)
- death of kidney tissue (possible kidney failure)
- blood in the urine
- broken bone(s)
- bone destruction (especially the legs, hips, and jaws)

- inflammation/swelling in or around the eyes (possible vision problems)
- blurry vision
- lung inflammation (possible difficulty breathing)
- difficulty breathing due to narrowing of the airways
- worsening of existing asthma
- allergic reaction, possibly life-threatening (such as difficulty breathing, low blood pressure, and/or organ failure)
- flu-like illness

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

## Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

During the **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

**CT scans** send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss** 

**of confidentiality**. Your data will be de-identified (all identifying information removed) during this study. The de-identified data will be stored in a password-protected, encrypted computer. The study doctor and members of the study team will have access to this data and the key linking you to your data. The data will be stored indefinitely (without time limit).

This study may involve unpredictable risks to the participants.

## **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant or breastfeed a baby while on this study.

If you can become pregnant and are sexually active, you must use at least 1 highly effective method of birth control while you are on study and for at least 90 days after you stop the study drugs. Talk to the study doctor about acceptable methods of birth control to use during the study.

If your partner is male and can father a child, they must use a condom while you are in the study and for 90 days after your last dose of study drugs.

If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

## **OPTIONAL PROCEDURES FOR THE STUDY**

**Optional Procedure #1:** If you agree, you will have a tumor biopsy at the time of progression (meaning the disease has gotten worse) or at the end-of-treatment visit for research testing related to your immune system and to learn if there have been any changes to the disease.

You do not have to agree to the optional procedure in order to take part in this study. There are no benefits to you for taking part in the optional procedure. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedure.

## **Optional Procedure Risks**

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

#### CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to have a biopsy if the disease progresses or at the end-of-treatment visit?

YES NO

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or Gateway for Cancer Research for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

## **Additional Information**

- 4. You may ask the study chair (Dr. Shannon Westin, at 713-794-4314) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this

study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. This is important because it may be dangerous or harmful to your health to suddenly stop taking the study drugs (stopping "cold turkey"). The study doctor will ask you to return to the clinic to complete the end-of-treatment visit, and may ask you to complete the follow-up visits, to check on your health. If you withdraw from this study, you can still choose to be treated at MD Anderson.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Gateway for Cancer Research, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: Gateway for Cancer Research.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

#### **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and Gateway for Cancer Research and/or shared with other researchers and/or institutions for use in future research.

## **Samples**

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research. Leftover samples will not be stored by Gateway for Cancer Research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples

#### **Genetic Research**

Samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you.

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

## **Authorization for Use and Disclosure of Protected Health Information (PHI):**

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson

- Gateway Foundation for Cancer Research, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study
- Study monitors and auditors who verify the accuracy of the information
- Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected. If you withdraw from the study, the study staff may ask if they can continue collecting the results of routine care from your medical record.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

| consent form for this study, or have had it read to it, ask questions, and talk about it with others as not o enroll me on this study. By signing this consent legal rights. I will be given a signed copy of this consent | needed. I give the study chair permission at form, I am not giving up any of my |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | _ |
| LEGALLY AUTHORIZED REPRESENTATIVE (L. The following signature line should only be filled out capacity to legally consent to take part in the study own behalf. | ut when the participant does not have the |
| SIGNATURE OF LAR | DATE |
| PRINTED NAME and RELATIONSHIP TO PARTIC | ICIPANT |
| WITNESS TO CONSENT I was present during the explanation of the researce 2021-0694. | rch to be performed under <b>Protocol</b> |
| SIGNATURE OF WITNESS TO THE VERBAL CO<br>PRESENTATION (OTHER THAN PHYSICIAN OF<br>A witness signature is only required for vulnerable adult part | R STUDY CHAIR) |
| PRINTED NAME OF WITNESS TO THE VERBAL | L CONSENT |
| PERSON OBTAINING CONSENT I have discussed this research study with the particepresentative, using language that is understandative fully informed this participant of the nature of risks and that the participant understood this explain | lable and appropriate. I believe that I of this study and its possible benefits and |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CON | <br>ISENT |

Protocol 2021-0694 June 29, 2022 Page 17 of 17

| TRANSLATOR |
|---|
| I have translated the above informed consent as written (without additions or subtractions) intoand assisted the people |
| (Name of Language) obtaining and providing consent by translating all questions and responses during the consent process for this participant. |
| NAME OF TRANSLATOR SIGNATURE OF TRANSLATOR DATE |
| ☐ Please check here if the translator was a member of the research team. (If checked, a witness, other than the translator, must sign the witness line below.) |
| SIGNATURE OF WITNESS TO THE VERBAL TRANSLATION (OTHER THAN TRANSLATOR, PARENT/GUARDIAN, OR STUDY CHAIR) |
| PRINTED NAME OF WITNESS TO THE VERBAL TRANSLATION |